CLINICAL TRIAL: NCT02040922
Title: An Observational Study of the Role of Antibiotics, Inflammation and Changes in Microbiota in the Development of Post-infective Bowel Dysfunction Following Infection With Campylobacter Jejuni or Coli
Brief Title: Campylobacter Enteritis and Post-Infective Bowel Dysfunction (PI-BD): Role of Antibiotics and Microbiota
Acronym: CERAMIC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other); Department of Health, United Kingdom (Other Government); King's College London (Other); University of Helsinki (Other)
Responsible Party: Sponsor
Other Study IDs: 13091; 13/EM/0310 (Other: National Research Ethics Committee)
Record Dates: First submitted 2014-01-14; First posted 2014-01-20 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Campylobacter Infections; Irritable Bowel Syndrome
Keywords: Antibiotics; Campylobacter; Diarrhoea; Enteritis; Microbiota; Calprotectin
MeSH Terms: conditions — Campylobacter Infections; Irritable Bowel Syndrome; Diarrhea; Enteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool (Faeces) Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post-Campylobacter: Adults with symptoms of intestinal infection who submit a stool sample from which Campylobacter jejuni or coli is cultured

SUMMARY:
The principal research objective is to determine the impact of antibiotic use on the risk of developing long term bowel symptoms after infection with the germ Campylobacter.

DETAILED DESCRIPTION:
The secondary research objectives are:

* To investigate how the particular strain of the Campylobacter germ that causes the infection, and the strength of the immune response that it stimulates in the bowel, affect the risk of long term bowel symptoms.
* To explore what changes occur after Campylobacter infection in the bacteria that usually live in the large bowel (microbiota) and the chemicals that they produce (short-chain fatty acids) when they digest nutrients. We will look for differences between people who recover fully and people who have long term bowel symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Clinical syndrome suggestive of intestinal infection, including symptoms such as new onset of abdominal pain, vomiting, diarrhoea, blood in stools, fever
* Submission of stool sample to Nottingham University Hospitals Microbiology Laboratory for investigation of these symptoms
* Campylobacter sp. cultured by selective media (standard clinical practice) from this stool sample

Exclusion Criteria:

* Pregnancy declared by the candidate
* History declared by the candidate of pre-existing gastrointestinal disorder, including but not limited to:

  * Inflammatory Bowel Disease
  * Coeliac Disease
  * Pancreatitis
  * Gallstone disease (biliary colic, cholecystitis)
  * Diverticulitis
  * Cancer of the gastrointestinal tract
  * Irritable Bowel Syndrome
* Reported history of previous resection of any part of the gastrointestinal tract other than appendix or gallbladder
* Intestinal stoma
* Habitual use of opiate analgesics likely to alter bowel function e.g. morphine
* Use of antibiotics in the preceding four weeks other than for treatment of index infection.
* Use of purgative products/ high dose laxatives for bowel preparation in the four weeks prior to index infection.
* Any condition where the candidate is likely to require a course of antibiotics in the next 3 months e.g. severe chronic respiratory disease, recurrent urinary tract infection, lower limb ulceration
* Inability to complete the symptom questionnaires e.g. cognitive dysfunction limiting memory and understanding
* Declared participation in any medical trials in the past 3 months
* Anyone who in the opinion of the investigator is unlikely to be able to comply with the protocol e.g. cognitive dysfunction, chaotic lifestyle related to substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults in the Nottinghamshire area with no previous history of gastrointestinal disorder or surgical resection. Those who submit a stoo lsample from which Campylobacter spp. is cultured will be invited to take part.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-02 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Yes/ no: Post-Infective bowel dysfunction (PI-BD) | 12 weeks after microbiological diagnosis of infection
  This will be defined by response to the question "have your bowels returned to normal since your Campylobacter infection?"

SECONDARY OUTCOMES:
Yes/ No: Post-Infective irritable bowel syndrome (PI-IBS) | 12 weeks after microbiological diagnosis of infection
  Symptoms meeting Rome III criteria for Irritable Bowel Syndrome (other than 6 month duration)

CONTACTS AND LOCATIONS:
Overall Officials: Robin C Spiller, MSc MD FRCP, Study Chair — University of Nottingham; Giles AD Major, BM BCh MRCP, Principal Investigator — University of Nottingham; Mathew Diggle, MSc PhD, Study Director — Nottingham University Hospitals NHS Trust; Richard Puleston, MBBS PhD, Study Director — University of Nottingham; Miranda Lomer, PhD RD, Study Director — King's College London
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jalanka J, Gunn D, Singh G, Krishnasamy S, Lingaya M, Crispie F, Finnegan L, Cotter P, James L, Nowak A, Major G, Spiller RC. Postinfective bowel dysfunction following Campylobacter enteritis is characterised by reduced microbiota diversity and impaired microbiota recovery. Gut. 2023 Mar;72(3):451-459. doi: 10.1136/gutjnl-2021-326828. Epub 2022 Sep 28. PMID 36171082
- See also: Departmental website — http://www.nddcbru.org.uk